CLINICAL TRIAL: NCT05713812
Title: "EFFECTS OF KINESIO-TAPING ON PAIN, POSTURAL STABILITY AND FUNCTION IN PERSONS WITH DISCOGENIC LOW BACK PAIN"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/4
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): * IFC + Hot pack for 20 minutes
  * MDT (prone positioning) for 10 minutes.
  * Lumbar SNAGs + lumbar rotation mobilization.
  * Home exercise plan: MDT for 10 min + patient education to avoid flexion based activities.
  * Sham Kinesiotape will be applied
  Interventions: Procedure: Control Treatment
- Experimental Group (Experimental): * IFC + Hot pack for 20 minutes
  * MDT (Prone positioning) for 10 minutes.
  * Lumbar SNAGs + lumbar rotation mobilization.
  * Home exercise plan: MDT for 10 min + patient education to avoid flexion based activities.
  * Kinesiotape will be applied
  Interventions: Procedure: Kinesiotaping

INTERVENTIONS:
Procedure: Kinesiotaping — Kinesiotape will be applied
  Arms: Experimental Group
Procedure: Control Treatment — IFC + Hot pack for 20 minutes MDT (prone positioning) for 10 minutes. Lumbar SNAGs + lumbar rotation mobilization. Home exercise plan: MDT for 10 min + patient education to avoid flexion based activities.
  Arms: Active Comparator

SUMMARY:
Low back pain is the leading cause of disability worldwide, the prevalence of low back pain can be as high as 43%. Past research has shown the positive effects of Kinesio taping in patients with chronic and nonspecific low back pain in pain reduction, improvement in postural stability, and improvement in function. However, no study has yet evaluated the effects of KT in persons with discogenic LBP. If found to be effective KT can be prescribed as a conservative & cost-effective treatment for patients with discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age20-45 years.
* Positive straight leg raise (SLR)
* Posterolateral disc bulge, herniation or prolapse indicated by MRI.
* Positive centralization and peripheralization phenomenon.

Exclusion Criteria:

* Participants having spondylolisthesis, fractures, tumors, osteoporosis, infection, or spinal stenosis.
* History of lumbar spine surgery and patients that are already receiving any physical therapy or exercise
* Skin allergy or sensitivity to the tape.
* Neurological, rheumatologic, or psychiatric disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Back Pain | 2 weeks.
  Back Pain will be measured via numerical pain rating scale. A higher score signifies greater pain.
Postural Stability | 2 weeks.
  Postural Stability will be measured via Biodex Balance System. A higher score signifies poorer stability.
Disability | 2 weeks.
  Disability will be measured via Oswestry Disability Index. A higher score signifies poorer outcome.
Gait velocity | 2 weeks.
  velocity of gait will be measured via gait analysis.
Stride length | 2 weeks.
  Stride length of gait will be measured via gait analysis.
Cadence | 2 weeks.
  Cadence of gait will be measured via gait analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sameen Tariq, DPT, Principal Investigator — Foundation University Islamabad; Muhammad Osama, PhD*, Study Director — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No